CLINICAL TRIAL: NCT03842865
Title: An Expanded Access Trial of Vigil (Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Immunotherapy) in Advanced Solid Tumors
Brief Title: Expanded Access of Vigil in Solid Tumors
Status: Temporarily not available | Type: Expanded Access
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-PTL-132
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor; Ewing Sarcoma; Ewing's Tumor Metastatic; Ewing's Sarcoma Metastatic; Advanced Gynecological Cancers; Ovarian Cancer; Cervical Cancer; Uterine Cancer
Keywords: Immunotherapy
MeSH Terms: conditions — Sarcoma, Ewing; Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — FANG vaccine

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: Vigil — Vigil is composed of autologous tumor cells harvested from the patient at the time of initial de-bulking surgery which are then transfected extracorporeally, with a plasmid encoding for the gene for GM-CSF, an immune-stimulatory cytokine, and a bifunctional, short hairpin RNA which specifically knocks down the expression of furin, the critical convertase responsible for production of the two TGβ isoforms (TGFβ-1 and TGFβ-2).
  Other Names: Engineered Autologous Tumor Cell Immunotherapy; FANG; IND 14205

SUMMARY:
This is an expanded access study involving an investigational product named Vigil. Vigil is considered immunotherapy. Patients who participated in another clinical trial sponsored by Gradalis, and had Vigil made from their tumor tissue removed from a standard operation, however failed the criteria to enroll in the other clinical trial to receive Vigil are eligible to screen for this expanded access trial to receive the Vigil made from their cancer cells.

In this study, eligible participants will receive intradermal (under the skin) injections of Vigil, once every 4 weeks (28 days) for 1-12 doses, depending on the number of doses that was made from the cancer cells and if the participant is clinically stable. During the treatment portion of the study, in addition to receiving Vigil injections, participants will also have a physical exam, blood collection for routine and research tests, and assessment of medications, adverse events, and performance status information will be collected. Radiological tumor assessments will be performed every 3 months from Cycle 1. Once treatment ends, participants will continue to be seen in the clinic every 3 months for similar assessments until disease progression occurs. After disease progression, participants will be contacted by phone 4 times a year to determine post study treatment and survival status information.

DETAILED DESCRIPTION:
This is an Expanded Access trial of Vigil (bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Immunotherapy) in Advanced Solid Tumors. Approximately 40 subjects who had tissue procured and Vigil manufactured but fail manufacturing release criteria under a previous Gradalis protocol are considered for this study.

Eligible participants will receive a minimum of 1 and a maximum of 12 doses of Vigil intradermal injections every 4 weeks as monotherapy. Participants will be managed in an outpatient setting. Hematologic function, liver enzymes, renal function and electrolytes will be monitored. Blood for immune function analyses in response to autologous tumor antigens will be collected at screening, Day 1 (prior to Vigil administration) at Cycles 2, 4, and 6, end of treatment (EOT); 3 months after EOT, and every 6 months thereafter for those in response follow up. For subjects with Ewing's sarcoma, blood for ctDNA analysis will be collected at screening, on Day 1 prior to Vigil administration at Cycles 2, 3, 4, and 6, and EOT.

ELIGIBILITY:
Study Enrollment Inclusion Criteria:

1. Histologically confirmed advanced or metastatic non-curable solid tumor.
2. Completed manufacture of at least 1 vial of Vigil, but failure of one or more manufacturing release criteria.
3. ECOG performance status (PS) 0-1 or Karnofsky performance status (KPS) / Lansky performance status (LS)≥ 70%.
4. Normal organ and marrow function as defined below:

   Absolute granulocyte count ≥1,000/mm3, Absolute lymphocyte count ≥400/mm3, Platelets ≥75,000/mm3, Hemoglobin ≥ 8.0 mg/dL, Total bilirubin ≤ institutional upper limit of normal*, AST(SGOT)/ALT(SGPT) ≤2x institutional upper limit of normal, Creatinine <1.5 mg/dL

   *documented Gilbert's syndrome may be considered after medical monitor review
5. No systemic therapy, immunologic therapy or investigational therapy within 2 weeks and no radiation therapy within 1 week prior to enrollment.
6. Subject has recovered to CTCAE Grade 1 (except for parameters noted in Item 4, above) or better from all adverse events associated with prior therapy or surgery. Pre-existing motor, sensory neurologic pathology or symptoms, or dermatologic toxicities must be recovered to CTCAE Grade 2 or better.
7. If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry.
8. Ability to understand and the willingness to sign a written informed protocol specific consent or a parental/guardian informed consent and pediatric assent when appropriate.

Study Enrollment Exclusion Criteria:

1. Medical condition requiring any form of chronic systemic immunosuppressive therapy (steroid or other) except physiologic replacement doses of hydrocortisone or equivalent (no more than 30 mg hydrocortisone or 10 mg prednisone equivalent daily) for < 30 days duration.
2. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
3. Receipt of greater than 2 lines of systemic treatment between Vigil manufacture and screening for this protocol.
4. Live vaccine used for the prevention of infectious disease administered < 30 days prior to the start of study therapy.
5. Post-surgery complication that in the opinion of the treating investigator would interfere with the subject's study participation or make it not in the best interest of the patient to participate.
6. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months.
7. Any documented history of autoimmune disease with exception of Type 1 diabetes on stable insulin regimen, hypothyroidism on stable dose of replacement thyroid medication, vitiligo, or asthma not requiring systemic steroids.
8. Known HIV or chronic Hepatitis B or C infection.
9. Known history of allergies or sensitivities to gentamicin.
10. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Study Director — Gradalis, Inc.
Locations (1):
- Texas Oncology - Pediatrics, Dallas, Texas, United States

REFERENCES:
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Background] Ghisoli M, Rutledge M, Stephens PJ, Mennel R, Barve M, Manley M, Oliai BR, Murphy KM, Manning L, Gutierrez B, Rangadass P, Walker A, Wang Z, Rao D, Adams N, Wallraven G, Senzer N, Nemunaitis J. Case Report: Immune-mediated Complete Response in a Patient With Recurrent Advanced Ewing Sarcoma (EWS) After Vigil Immunotherapy. J Pediatr Hematol Oncol. 2017 May;39(4):e183-e186. doi: 10.1097/MPH.0000000000000822. PMID 28338569
- [Background] Oh J, Barve M, Matthews CM, Koon EC, Heffernan TP, Fine B, Grosen E, Bergman MK, Fleming EL, DeMars LR, West L, Spitz DL, Goodman H, Hancock KC, Wallraven G, Kumar P, Bognar E, Manning L, Pappen BO, Adams N, Senzer N, Nemunaitis J. Phase II study of Vigil(R) DNA engineered immunotherapy as maintenance in advanced stage ovarian cancer. Gynecol Oncol. 2016 Dec;143(3):504-510. doi: 10.1016/j.ygyno.2016.09.018. Epub 2016 Sep 24. PMID 27678295
- [Background] Rocconi RP, Grosen EA, Ghamande SA, Chan JK, Barve MA, Oh J, Tewari D, Morris PC, Stevens EE, Bottsford-Miller JN, Tang M, Aaron P, Stanbery L, Horvath S, Wallraven G, Bognar E, Manning L, Nemunaitis J, Shanahan D, Slomovitz BM, Herzog TJ, Monk BJ, Coleman RL. Gemogenovatucel-T (Vigil) immunotherapy as maintenance in frontline stage III/IV ovarian cancer (VITAL): a randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Oncol. 2020 Dec;21(12):1661-1672. doi: 10.1016/S1470-2045(20)30533-7. PMID 33271095
- [Background] Oh J, Barve M, Senzer N, Aaron P, Manning L, Wallraven G, Bognar E, Stanbery L, Horvath S, Manley M, Nemunaitis J, Walter A, Rocconi RP. Long-term follow-up of Phase 2A trial results involving advanced ovarian cancer patients treated with Vigil(R) in frontline maintenance. Gynecol Oncol Rep. 2020 Sep 17;34:100648. doi: 10.1016/j.gore.2020.100648. eCollection 2020 Nov. No abstract available. PMID 33364285